CLINICAL TRIAL: NCT06798376
Title: The Comparison of Different Cycles of PD-1 Blockades Combined with Chemotherapy As Neoadjuvant Therapy for Patients with Advanced Gastric Cancer
Brief Title: Different Cycles of Neoadjuvant PD-1 Blockades + Chemotherapy for Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xinxin Wang, Prof., Chinese PLA General Hospital
Other Study IDs: S2024-823
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gastric Adenocarcinoma
Keywords: Advanced Gastric Adenocarcinoma; Neoadjuvant; Immunotherapy; Chemotherapy; Cycles
MeSH Terms: interventions — Drug Therapy; Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: The group A contains participants who received ≤4 cycles of neoadjuvant PD-1 inhibitor combined with chemotherapy and then received gastrectomy.
  Interventions: Drug: ≤4 cycles of neoadjuvant PD-1 Inhibitors combined with chemotherapy; Procedure: Gastrectomy
- Group B: The group B contains participants who received ≥5 cycles of neoadjuvant PD-1 inhibitor combined with chemotherapy and then received gastrectomy.
  Interventions: Drug: ≥5 cycles of neoadjuvant PD-1 Inhibitors combined with chemotherapy; Procedure: Gastrectomy

INTERVENTIONS:
Drug: ≤4 cycles of neoadjuvant PD-1 Inhibitors combined with chemotherapy — Any PD-1 inhibitors combined with any chemotherapy regimen given before surgery for no more than 4 cycles
  Groups: Group A
Drug: ≥5 cycles of neoadjuvant PD-1 Inhibitors combined with chemotherapy — Any PD-1 inhibitors combined with any chemotherapy regimen given before surgery for no less than 5 cycles
  Groups: Group B
Procedure: Gastrectomy — Any type of surgical procedure for gastric adenocarcinoma patients in which part or all of the stomach is removed

SUMMARY:
The goal of this observational study is to analyze the impact of different durations of neoadjuvant PD-1 inhibitor combined with chemotherapy on tumor regression and safety in patients with advanced gastric cancer. The main questions it aims to answer are:

* Does the duration of neoadjuvant treatment influence tumor regression grading (TRG)?
* How does treatment duration affect perioperative safety and clinical outcomes?

Participants who have previously undergone neoadjuvant PD-1 inhibitor combined with chemotherapy followed by surgery as part of their routine medical care will have their clinical data retrospectively reviewed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Non-bedridden patients aged 18-90 years;
* Histologically confirmed gastric or gastroesophageal junction adenocarcinoma by biopsy;
* Evaluated as resectable advanced gastric cancer via CT, MRI, or laparoscopic exploration;
* No prior anti-tumor treatments such as chemotherapy, radiotherapy, or immunotherapy;
* No history of other malignancies within the past 5 years;
* Received at least one cycle of PD-1 inhibitor combined with chemotherapy preoperatively, with no restrictions on the specific PD-1 inhibitor or chemotherapeutic agents;
* Underwent radical gastrectomy after neoadjuvant therapy;
* No severe underlying diseases.

Exclusion Criteria:

* Incomplete or inaccessible clinical and pathological data;
* Postoperative pathology confirming non-gastric or non-gastroesophageal junction adenocarcinoma;
* Distant metastases present prior to treatment;
* Concurrent diagnosis of other malignancies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer patients who received preoperative PD-1 inhibitor combined with chemotherapy and gastrectomy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Regression Grading (TRG) | Approximately 1 week after surgery (when the pathology examination report available)
  Tumor Regression Grading (TRG) based on the Chinese Society of Clinical Oncology (CSCO) guidelines ranging from 0 (no residual tumor) to 3 (extensive residual tumor cells with no or minimal tumor cell necrosis), with higher scores indicating worse outcomes

SECONDARY OUTCOMES:
Safety | From the start of neoadjuvant chemotherapy to 7 days after surgery
  Adverse events during neoadjuvant therapy and postoperative complications
R0 resection | Approximately 1 week after surgery (when the pathology examination report available)
  Complete removal of a tumor with no residual cancer cells at the surgical margins, confirmed by pathological examination
Operative time | On the day of the surgery (can be obtained immediately after the completion of the surgery)
  The total duration of a surgical procedure, measured from the first incision to the completion of wound closure
Time to first flatus | From date of surgery until the date of first flatus, assessed up to 10 days post-surgery
  The duration from the completion of surgery to the first passing of gas (flatus) by the patient
Nutritional Risk Screening 2002 (NRS 2002) | Approximately 1 week after completing all neoadjuvant therapy
  The Nutritional Risk Screening 2002 (NRS 2002) is a scale used to assess the nutritional risk of hospitalized patients. The score ranges from 0 to 7, with higher scores indicating a higher risk of malnutrition. A score of 0 signifies no nutritional risk, while a score of 3 or higher indicates a significant nutritional risk that may require intervention.
YpTNM staging | Approximately 1 week after surgery (when the pathology examination report available)
  Pathological classification used to assess cancer characteristics after neoadjuvant therapy, based on the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition.
Dissected lymph node number | Approximately 1 week after surgery (when the pathology examination report available)
  The total number of lymph nodes surgically removed and examined
Positive lymph node number | Approximately 1 week after surgery (when the pathology examination report available)
  The number of lymph nodes found to contain cancer cells upon pathological examination

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study containing data related to the outcomes observed in the study, without any personal information or other data of the patients will be shared.
Time Frame: Within 3 years after the publication of the study results
Access Criteria: The datasets used and/or analyzed during the current study containing data related to the outcomes observed in the study, without any personal information or other data of the patients will be shared. Qualified medical professionals can access the datasets by submitting a written request and obtaining approval from the principal investigator and other researchers involved in the study.

REFERENCES:
- [Background] Hayashi T, Yoshikawa T, Sakamaki K, Nishikawa K, Fujitani K, Tanabe K, Misawa K, Matsui T, Miki A, Nemoto H, Fukunaga T, Kimura Y, Hihara J. Primary results of a randomized two-by-two factorial phase II trial comparing neoadjuvant chemotherapy with two and four courses of cisplatin/S-1 and docetaxel/cisplatin/S-1 as neoadjuvant chemotherapy for advanced gastric cancer. Ann Gastroenterol Surg. 2020 Jul 16;4(5):540-548. doi: 10.1002/ags3.12352. eCollection 2020 Sep. PMID 33005849
- [Background] Yoshikawa T, Tanabe K, Nishikawa K, Ito Y, Matsui T, Kimura Y, Hirabayashi N, Mikata S, Iwahashi M, Fukushima R, Takiguchi N, Miyashiro I, Morita S, Miyashita Y, Tsuburaya A, Sakamoto J. Induction of a pathological complete response by four courses of neoadjuvant chemotherapy for gastric cancer: early results of the randomized phase II COMPASS trial. Ann Surg Oncol. 2014 Jan;21(1):213-9. doi: 10.1245/s10434-013-3055-x. Epub 2013 Jul 10. PMID 23838904
- [Background] Lorenzen S, Gotze TO, Thuss-Patience P, Biebl M, Homann N, Schenk M, Lindig U, Heuer V, Kretzschmar A, Goekkurt E, Haag GM, Riera-Knorrenschild J, Bolling C, Hofheinz RD, Zhan T, Angermeier S, Ettrich TJ, Siebenhuener AR, Elshafei M, Bechstein WO, Gaiser T, Loose M, Sookthai D, Kopp C, Pauligk C, Al-Batran SE; AIO and SAKK Study Working Groups. Perioperative Atezolizumab Plus Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel for Resectable Esophagogastric Cancer: Interim Results From the Randomized, Multicenter, Phase II/III DANTE/IKF-s633 Trial. J Clin Oncol. 2024 Feb 1;42(4):410-420. doi: 10.1200/JCO.23.00975. Epub 2023 Nov 14. PMID 37963317
- [Background] Sun W, Veeramachaneni N, Al-Rajabi R, Madan R, Kasi A, Al-Kasspooles M, Baranda J, Saeed A, Phadnis MA, Godwin AK, Olyaee M, Streeter N, Nagji A, Dai J, Williamson S. A phase II study of perioperative pembrolizumab plus mFOLFOX in patients with potentially resectable esophagus, gastroesophageal junction (GEJ), and stomach adenocarcinoma. Cancer Med. 2023 Aug;12(15):16098-16107. doi: 10.1002/cam4.6263. Epub 2023 Jun 16. PMID 37326317
- [Background] Yuan SQ, Nie RC, Jin Y, Liang CC, Li YF, Jian R, Sun XW, Chen YB, Guan WL, Wang ZX, Qiu HB, Wang W, Chen S, Zhang DS, Ling YH, Xi SY, Cai MY, Huang CY, Yang QX, Liu ZM, Guan YX, Chen YM, Li JB, Tang XW, Peng JS, Zhou ZW, Xu RH, Wang F. Perioperative toripalimab and chemotherapy in locally advanced gastric or gastro-esophageal junction cancer: a randomized phase 2 trial. Nat Med. 2024 Feb;30(2):552-559. doi: 10.1038/s41591-023-02721-w. Epub 2024 Jan 2. PMID 38167937
- [Background] Raimondi A, Lonardi S, Murgioni S, Cardellino GG, Tamberi S, Strippoli A, Palermo F, De Manzoni G, Bencivenga M, Bittoni A, Chiodoni C, Lorenzini D, Todoerti K, Manca P, Sangaletti S, Prisciandaro M, Randon G, Nichetti F, Bergamo F, Brich S, Belfiore A, Bertolotti A, Stetco D, Guidi A, Torelli T, Vingiani A, Joshi RP, Khoshdeli M, Beaubier N, Stumpe MC, Nappo F, Leone AG, Pircher CC, Leoncini G, Sabella G, Airo' Farulla L, Alessi A, Morano F, Martinetti A, Niger M, Fassan M, Di Maio M, Kaneva K, Milione M, Nimeiri H, Sposito C, Agnelli L, Mazzaferro V, Di Bartolomeo M, Pietrantonio F. Tremelimumab and durvalumab as neoadjuvant or non-operative management strategy of patients with microsatellite instability-high resectable gastric or gastroesophageal junction adenocarcinoma: the INFINITY study by GONO. Ann Oncol. 2025 Mar;36(3):285-296. doi: 10.1016/j.annonc.2024.11.016. Epub 2024 Dec 3. PMID 39637944
- [Background] Andre T, Tougeron D, Piessen G, de la Fouchardiere C, Louvet C, Adenis A, Jary M, Tournigand C, Aparicio T, Desrame J, Lievre A, Garcia-Larnicol ML, Pudlarz T, Cohen R, Memmi S, Vernerey D, Henriques J, Lefevre JH, Svrcek M. Neoadjuvant Nivolumab Plus Ipilimumab and Adjuvant Nivolumab in Localized Deficient Mismatch Repair/Microsatellite Instability-High Gastric or Esophagogastric Junction Adenocarcinoma: The GERCOR NEONIPIGA Phase II Study. J Clin Oncol. 2023 Jan 10;41(2):255-265. doi: 10.1200/JCO.22.00686. Epub 2022 Aug 15. PMID 35969830
- [Background] Rha SY, Oh DY, Yanez P, Bai Y, Ryu MH, Lee J, Rivera F, Alves GV, Garrido M, Shiu KK, Fernandez MG, Li J, Lowery MA, Cil T, Cruz FM, Qin S, Luo S, Pan H, Wainberg ZA, Yin L, Bordia S, Bhagia P, Wyrwicz LS; KEYNOTE-859 investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for HER2-negative advanced gastric cancer (KEYNOTE-859): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Nov;24(11):1181-1195. doi: 10.1016/S1470-2045(23)00515-6. Epub 2023 Oct 21. PMID 37875143
- [Background] Qiu MZ, Oh DY, Kato K, Arkenau T, Tabernero J, Correa MC, Zimina AV, Bai Y, Shi J, Lee KW, Wang J, Poddubskaya E, Pan H, Rha SY, Zhang R, Hirano H, Spigel D, Yamaguchi K, Chao Y, Wyrwicz L, Disel U, Cid RP, Fornaro L, Evesque L, Wang H, Xu Y, Li J, Sheng T, Yang S, Li L, Moehler M, Xu RH; RATIONALE-305 Investigators. Tislelizumab plus chemotherapy versus placebo plus chemotherapy as first line treatment for advanced gastric or gastro-oesophageal junction adenocarcinoma: RATIONALE-305 randomised, double blind, phase 3 trial. BMJ. 2024 May 28;385:e078876. doi: 10.1136/bmj-2023-078876. PMID 38806195
- [Background] Xu J, Jiang H, Pan Y, Gu K, Cang S, Han L, Shu Y, Li J, Zhao J, Pan H, Luo S, Qin Y, Guo Q, Bai Y, Ling Y, Yang J, Yan Z, Yang L, Tang Y, He Y, Zhang L, Liang X, Niu Z, Zhang J, Mao Y, Guo Y, Peng B, Li Z, Liu Y, Wang Y, Zhou H; ORIENT-16 Investigators. Sintilimab Plus Chemotherapy for Unresectable Gastric or Gastroesophageal Junction Cancer: The ORIENT-16 Randomized Clinical Trial. JAMA. 2023 Dec 5;330(21):2064-2074. doi: 10.1001/jama.2023.19918. PMID 38051328
- [Background] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Wu X, Gu Z, Chen Y, Chen B, Chen W, Weng L, Liu X. Application of PD-1 Blockade in Cancer Immunotherapy. Comput Struct Biotechnol J. 2019 May 23;17:661-674. doi: 10.1016/j.csbj.2019.03.006. eCollection 2019. PMID 31205619
- [Background] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Background] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751